CLINICAL TRIAL: NCT04373356
Title: Non-invasive and Minimal Intervention in Dental Caries Management: Randomized Clinical Study
Brief Title: Non-invasive Caries Management: Clinical Study
Acronym: NICM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 115761
Record Dates: First submitted 2020-04-28; First posted 2020-05-04 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Caries,Dental; Caries Arrested
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resin Infiltration (Experimental): The interproximal surface with initial dental caries that are selected for this group will be treated using the resin infiltration ICON (DMG, Germany) and 5% Sodium Fluoride Varnish
  Interventions: Device: Resin Infiltration
- Sodium Fluoride Varnish (Active Comparator): The interproximal surface with initial dental caries that are selected for this group will be treated using topical application of 5% Sodium Fluoride Varnish.
  Interventions: Device: Sodium Fluoride Varnish

INTERVENTIONS:
Device: Resin Infiltration — Patients will be instructed about enhancing their oral hygiene, and will be asked to brush their teeth twice a day with fluoride toothpaste, and use dental floss daily. In short, teeth will be isolated with a rubber dam and ICON will be applied following the manufacturer's instructions. After that, the rubber dam will be removed and 5% NaF Varnish will be applied.
  Standardized digital bitewing radiograph will be taken at baseline and one year after treatment for caries lesion progression comparison.
  Arms: Resin Infiltration
Device: Sodium Fluoride Varnish — Patients will be instructed about enhancing their oral hygiene, and will be asked to brush their teeth twice a day with fluoride toothpaste, and use dental floss daily. In short, teeth will be isolated with cotton roll and 5% NaF varnish will be applied following the manufacturer's instructions.
  Standardized digital bitewing radiograph will be taken at baseline and one year after treatment for caries lesion progression comparison.
  Arms: Sodium Fluoride Varnish

SUMMARY:
Clinical trial to compare non-invasive and minimally-invasive therapies on the progression of the caries lesions. Clinical investigation of resin infiltration versus sodium fluoride (5% NaF) varnish application.

DETAILED DESCRIPTION:
Dental caries is the most globally prevalent disease that affects thousands of adults and children. Caries is a biofilm-mediated, sugar-driven, multifactorial, and dynamic disease that results from the imbalance between demineralization and remineralization of the dental hard tissues. Preventing the onset of the disease should be the primary goal; however, once the disease is present efforts should be made by both patient and clinician to successfully reestablish the mineralization balance by the use of preventive and/or minimally-invasive methods when possible. The sodium fluoride (5% NaF) varnish is one of the most common therapies used as a non-invasive approach for caries prevention and remineralization; and, the resin infiltration materials are indicated for the minimal intervention of non-cavitated occlusal and proximal caries. The minimal intervention has been considered the new concept of caries management. Although several studies discussing minimal intervention or non-intervention are available, there is a lack of published randomized controlled trials (RCTs) providing data about the use of non-invasive therapies on incipient lesions, and its correlation with the patient's caries risk. The aim of this study is to evaluate the efficacy non-invasive and minimally-invasive therapies on the progression of the caries lesions considering the patient's caries risk.

This study will be conducted in the province of Ontario, Canada. A total of thirty patients (15 to 50 years old), who present with a minimum of two incipient proximal carious lesions on the proximal surfaces of posterior teeth (non-cavitated lesions identified as small, faint radiolucent areas seen on the intra-oral radiographs) will be asked to participate in this study. The radiologic assessment of incipient lesions will be performed by a dental radiologist, blinded to the selected treatment groups, by comparison of the radiographs imaging over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients must present at least two non-cavitated proximal caries lesions
* Patients must be able to give informed consent in English
* Patients must be resident in London, Ontario, or nearby locales with community fluoridation

Exclusion Criteria:

* Patients presenting proximal caries that are beyond the outer third of dentin
* Patients suffering from a disability that impairs dental hygiene performance
* Patients that are unable to perform her/his own oral hygiene

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Caries lesion progression | One year follow up
  Evaluate caries lesion progression after using DMG Icon-infiltrative resin and/or 5% NaF Varnish by comparison of baseline and one year post-treatment radiographics.

SECONDARY OUTCOMES:
Caries risk assessment | One year follow up
  Evaluate non-invasive and minimally-invasive therapies on the progression of the caries lesions correlated with the patient's caries risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Schulich School of Medicine & Dentistry - Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No